CLINICAL TRIAL: NCT04033237
Title: Project 4, Study 2: Extended Exposure to Low Nicotine Content Cigarettes in Pregnant Women
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency); University of Kentucky (Other)
Responsible Party: Principal Investigator, Sarah Heil, Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHRMS 16-390; U54DA036114 (NIH)
Record Dates: First submitted 2019-07-23; First posted 2019-07-26 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Tobacco Use Disorder
Keywords: Biomarkers of exposure; Compensatory smoking; Nicotine dependence; Reduced nicotine cigarettes; Tobacco withdrawal; Women; Pregnancy; Health disparities; Vulnerable populations
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Very low nicotine content cigarettes (Experimental)
  Interventions: Other: Very low nicotine content cigarettes
- Usual Brand (No Intervention)

INTERVENTIONS:
Other: Very low nicotine content cigarettes — Cigarettes containing 0.4 mg nicotine/g tobacco
  Arms: Very low nicotine content cigarettes

SUMMARY:
Study 2 will evaluate the effects of extended exposure to cigarettes with varying levels of nicotine in pregnant smokers who have less than an Associate's degree. This study will be limited to two conditions: usual brand vs. 0.4 mg nicotine/g tobacco. After a baseline period in which daily smoking rate and other baseline assessments are completed, participants will be randomly (by chance) assigned to either their usual brand or the very low nicotine content condition and followed for 12 weeks.

DETAILED DESCRIPTION:
Some inclusion/exclusion criteria are purposely omitted at this time to preserve scientific integrity. They will be included after the trial is complete.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ages 18-44 years
* Gestational age ≤ 25 weeks

Exclusion Criteria:

* Male
* Under 18 years old
* Over 44 years old
* Gestational age > 25 weeks

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah H. Heil, Principal Investigator — University of Vermont
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - University of Vermont, Burlington, Vermont

REFERENCES:
- [Derived] Heil SH, Kock LS, Harfmann RF, Ashford KB, Barnett J, McCubbin A, DeSarno MJ, Higgins ST. Pilot randomized clinical trial examining use of very low nicotine content cigarettes during pregnancy in the United States. Prev Med. 2025 Dec;201:108351. doi: 10.1016/j.ypmed.2025.108351. Epub 2025 Jul 5. PMID 40623557

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Brand: Participant's usual brand cigarettes
Period: Overall Study
Arm/Group | Very Low Nicotine Content Cigarettes | Usual Brand
Started | 16 | 14
Completed | 12 | 11
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Very Low Nicotine Content Cigarettes | Usual Brand | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.31 (4.80) | 27.57 (4.77) | 27.97 (4.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Latino White | 15 | 14 | 29
  Non-Latino other | 1 | 0 | 1
Gestational age at screening [Mean (Standard Deviation); unit: Weeks] | 11.94 (4.99) | 13.43 (6.26) | 12.63 (5.57)
Cigarettes per day pre-pregnancy [Mean (Standard Deviation); unit: Cigarettes per day] | 18.38 (5.91) | 23.93 (14.08) | 20.97 (10.72)
Cigarettes per day [Mean (Standard Deviation); unit: Cigarettes per day] | 19.19 (8.15) | 16.21 (8.05) | 17.80 (8.10)

OUTCOME MEASURES:

1. Primary Outcome: Total Cigarettes Per Day
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Cigarettes per day
Arm/Group | Very Low Nicotine Content Cigarettes | Usual Brand
Number analyzed (Participants) | 12 | 11
Cigarettes per day | 16.31 (2.63) | 18.36 (2.32)

ADVERSE EVENTS:
Time Frame: 12-week intervention period
Arm/Group | Very Low Nicotine Content Cigarettes | Usual Brand
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/14
Other Adverse Events (participants affected / at risk) | 11/16 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Very Low Nicotine Content Cigarettes (N=16) | Usual Brand (N=14)
Placenta previa (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Very Low Nicotine Content Cigarettes (N=16) | Usual Brand (N=14)
Cardiac disorders (Cardiac disorders) | 2 (2) | 0 (0)
Gastrointestinal disorders (Gastrointestinal disorders) | 4 (9) | 2 (2)
General disorder and administration (General disorders) | 3 (5) | 0 (0)
Infections and infestations (Infections and infestations) | 4 (4) | 2 (2)
Musculoskeletal and connective tissue (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Nervous system disorders (Nervous system disorders) | 1 (3) | 1 (1)
Pregnancy, puerperium and perinatal (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 3 (4)
Psychiatric disorders (Psychiatric disorders) | 2 (3) | 2 (2)
Respiratory, thoracic and mediastina (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Vascular disorders (Vascular disorders) | 2 (2) | 2 (2)
Breath carbon monoxide >50ppm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Breath carbon monoxide >100% baseline level (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cigarettes per day >/= 100% baseline level (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Increased Beck Depression Inventory score (Psychiatric disorders) | 7 (8) | 8 (11)
Increased Overall Anxiety Severity and Impairment Scale score (Psychiatric disorders) | 4 (5) | 5 (7)

LIMITATIONS AND CAVEATS:
The sample included participants who smoke more than is typical during pregnancy and the sample size (N=30) was small. Study generality may be limited by the high smoking rate and the small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/37/NCT04033237/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT04033237/SAP_001.pdf